CLINICAL TRIAL: NCT00349310
Title: Profile of Depressive Symptoms in Parkinson's Disease (PRODEST-PD)
Brief Title: Profile of Depressive Symptoms in Parkinsons Disease
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 248.597
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Parkinson Disease; Depression
MeSH Terms: conditions — Parkinson Disease; Depression | interventions — Pramipexole

INTERVENTIONS:
Drug: Pramipexole

SUMMARY:
To explore or establish the relationship between cognitive, mood and motor symptoms in PD to scores on depression rating scales in a naturalistic setting.

ELIGIBILITY:
Inclusion_Criteria:

Observation criteria:

* are able to provide written informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* have idiopathic Parkinsons disease according to the United Kingdom Parkinsons Disease Society Brain Bank Diagnostic Criteria for Parkinsons disease
* show no impairment of cognitive function (MMSE score ?24)
* are with or without symptoms of depression (full range)
* are stable on anti-Parkinson/anti-depressive treatment for at least 1 month before entering the study
* are or are not on concomitant antidepressant treatment
* are in the on state during the observation period
* did not previously undergo PD surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1018
Dates: Start 2006-04-01 (Actual); Primary Completion 2006-10-01 (Actual); Study Completion 2006-10-01 (Actual)

PRIMARY OUTCOMES:
HADS, HAMD-17, BDI-1A, FAB (cognitive), DSM-IV (mood- part A, B, C, E) and UPDRS | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim BV/Alkmaar
Locations (23):
- Austria (2):
  - Boehringer Ingelheim Investigational Site, Innsbruck
  - Boehringer Ingelheim Investigational Site, Vienna
- France (2):
  - Hopital Rangueil, Toulouse
  - Hopital Purpan, Toulouse
- Germany (6):
  - Neurologisches Fachkrankenhaus fur, Beelitz-Heilstätten
  - Universitatsklinikum Carl Gustav Carus Dresden, Dresden
  - Boehringer Ingelheim Investigational Site, Gera
  - Gertrudis-Kliniken Biskirchen, Leun
  - Boehringer Ingelheim Investigational Site, Unterhaching
  - Parkinson Klinik Wolfach, Wolfach
- Italy (4):
  - Policlinico di Catania, Catania
  - Azienda Ospedaliera S. Martino, Genova
  - Universita Federico II, Napoli
  - Universita La Sapienza di Roma, Roma
- Academisch Ziekenhuis Maastricht, Maastricht, Netherlands
- Spain (3):
  - Hospital de Cruces. Neurology, Baracaldo / Bilbao
  - Hospital Clinic i Provincial. Neurology, Barcelona
  - Hospital Puerta del Mar. Neurology, Cadiz
- Switzerland (3):
  - Clinica Hildebrand, Brissago
  - Hopital Cantonal (HUG), Geneva
  - Kantonsspital St. Gallen, Sankt Gallen
- United Kingdom (2):
  - Boehringer Ingelheim Investigational Site, London
  - Boehringer Ingelheim Investigational Site, Newark